CLINICAL TRIAL: NCT06928766
Title: Effects of Eszopiclone and Lemborexant in People With Obstructive Sleep Apnoea (OSA) With a Low Arousal Threshold Who Have Difficulty Maintaining or Falling Asleep (ELOSA): A Double-blind, Placebo-controlled, Randomised, Trial.
Brief Title: Effects of Eszopiclone and Lemborexant in People With OSA With a Low Arousal Threshold Who Have Difficulty Sleeping
Acronym: ELOSA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Flinders University (Other)
Responsible Party: Principal Investigator, Professor Danny Eckert, Director, Adelaide Institute for Sleep Health, Professor, College of Medicine and Public Health and Matthew Flinders Fellow, Flinders University, Flinders University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7849; 1196261 (Other Grant/Funding Number: National health and medical research council of Australia)
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: OSA - Obstructive Sleep Apnea
Keywords: sleep disordered breathing; arousal; COMISA
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Eszopiclone; Sugars; lemborexant

STUDY DESIGN:
Intervention Model Description: Oral capsules (Eszopiclone 3mg and lemborexant 10mg) taken together or placebo equivalent , order is randomized. After at least a week washout the opposite agent will be given.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Eszopiclone 3mg and lemborexant 10mg (Experimental): Both Eszopiclone 3mg and Lemborexant 10mg in the form of capsules taken before bedtime. Dosages is taken on one instance for one night only.
  Interventions: Drug: Eszopiclone 3 mg; Drug: Lemborexant 10mg
- Placebo (Placebo Comparator): Placebo capsules that look exactly like the study drugs, taken before bedtime. Dosage is taken on one instance for one night only.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eszopiclone 3 mg — Both eszopiclone and lemborexant taken together at bedtime for one night
  Other Names: Lunesta
  Arms: Eszopiclone 3mg and lemborexant 10mg
Drug: Placebo — Placebo sugar pills that looks like the eszopiclone and lemborexant capsules taken at bedtime for one night.
  Other Names: Sugar pill
  Arms: Placebo
Drug: Lemborexant 10mg — Both eszopiclone and lemborexant taken together at bedtime for one night
  Other Names: Dayvigo
  Arms: Eszopiclone 3mg and lemborexant 10mg

SUMMARY:
Insomnia and obstructive sleep apnoea (OSA) are very common conditions, collectively estimated to affect 2 billion people globally, and share many of the same symptoms. It is also common for people to have both insomnia and sleep apnoea (COMISA). Indeed, 30 to 40% of patients with chronic insomnia also fulfil the diagnostic criteria for OSA. These people can be particularly challenging to treat with conventional therapy approaches.

People get OSA for different reasons. One key cause is waking up too easily to minor airway narrowing episodes (a low arousal threshold).

Accordingly, this study aims to increase the arousal threshold using a combination approach with a GABAergic and an orexin agent in appropriately selected individuals (i.e., the clinically relevant group of people with OSA with a low arousal threshold and difficulty maintain or initiating sleep). Sleep, breathing and next day performance will be compared across two monitored overnight sleep studies (placebo vs the study drugs).

DETAILED DESCRIPTION:
Background:

Insomnia and obstructive sleep apnoea (OSA) are very common conditions, collectively estimated to affect 2 billion people globally, and share many of the same symptoms. It is also common for people to have both insomnia and sleep apnoea (COMISA). Indeed, 30 to 40% of patients with chronic insomnia also fulfil the diagnostic criteria for OSA. These people can be particularly challenging to treat with conventional therapy approaches.

OSA is characterised by repeated narrowing and closure of the upper airway during sleep, desaturation in oxygen levels, and fragmented sleep. OSA is a heterogeneous disease, with anatomical crowding of the upper airway and at least three distinct non-anatomical endotypes. The non-anatomical OSA endotypes include high loop gain (unstable control of breathing), poor upper airway dilator muscle function, and a low arousal threshold (ArTH- waking up too easily to minor airway narrowing events). Each OSA endotype represents a novel therapeutic target. Adding to the complexity of OSA, more than one endotype can contribute to a person's OSA. While the first line treatment for OSA, continuous positive airway pressure (CPAP) is efficacious, long-term compliance is only 40 to 70%. Those with a low ArTH endotype have markedly lower CPAP uptake and compliance.

Indeed, people with a low ArTH endotype experience frequent cortical arousals (awakenings) leading to fragmented and non-restorative sleep. Frequent cortical arousals prevent transitioning into deeper sleep states that are characterised by more stable breathing. Thus, strategies to increase the arousal threshold to stabilise breathing and reduce OSA severity in people who wake up easily (low ArTH) have been investigated as a novel therapeutic target. For example, commonly used hypnotic agents such as eszopiclone and trazodone can increase the arousal threshold and reduce OSA severity in people with a low ArTH. More recently, we have shown that 50mg quetiapine also improves sleep and reduces OSA severity in people with OSA who report difficulty maintaining sleep. However, the extent to which common hypnotic agents increase the arousal threshold in people with OSA is modest at best (~20%). This limits the therapeutic efficacy for people with OSA.

Orexin has been identified as an important sleep wake modulator. Accordingly, new orexin antagonists have been developed as novel sleep promotion aids for the treatment of insomnia. For example, the orexin antagonist, Lemborexant, has been shown to be safe and efficacious for the treatment of insomnia including in the elderly and people with OSA.

Given that current monotherapy approaches to increase the arousal threshold in people with OSA have only modestly increased the threshold for arousal with correspondingly modest reductions in OSA severity, there is a need to investigate the potential role for combination hypnotic therapy. Accordingly, this study aims to target two key sleep/wake mechanisms (the GABAergic and orexin systems) to determine if this combination approach yields greater therapeutic benefit than previous attempts with monotherapy in appropriately selected individuals (i.e., the clinically relevant group of people with OSA with a low ArTH and difficulty maintain or initiating sleep).

ELIGIBILITY:
Inclusion Criteria:

* Moderate or more difficulty "staying or initiating asleep" score on the Insomnia Severity Index questionnaire
* Obstructive Sleep Apnoea (OSA), Apnoea Hypopnea Index ≥ 10 events/hour
* Low arousal respiratory threshold OSA endotype
* BMI ≤35 kg/m2

Exclusion Criteria:

* Concomitant medications that interact or are contraindicated with eszopiclone, zopiclone, and Lemborexant
* Concomitant medications known to influence breathing, sleep, arousal, or muscle physiology
* Current pregnancy or breast-feeding
* Current or recent other medical conditions likely to affect results or safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in OSA severity (eszopiclone and lemborexant night vs. placebo night) | Two non-consecutive single night sleep studies (eszopiclone and lemborexant night vs. placebo night) up to one month apart.
  OSA severity as measured by the apnoea hypopnea index (units: number of respiratory events/h sleep) during overnight in-laboratory polysomnography.

SECONDARY OUTCOMES:
Change in nadir overnight hypoxemia (eszopiclone and lemborexant night vs. placebo night) | Two non-consecutive single night sleep studies (eszopiclone and lemborexant night vs. placebo night) up to one month apart.
  Nadir overnight oxygen saturation during sleep (units: %) measured via pulse oximetry during overnight in-laboratory polysomnography.
Change in mean overnight hypoxemia (eszopiclone and lemborexant night vs. placebo night) | Two non-consecutive single night sleep studies (eszopiclone and lemborexant night vs. placebo night) up to one month apart.
  Mean overnight oxygen saturation during sleep (units: %) measured via pulse oximetry during overnight in-laboratory polysomnography.
Change in time below 90% blood arterial oxygen saturation (eszopiclone and lemborexant night vs. placebo night) | Two non-consecutive single night sleep studies (eszopiclone and lemborexant night vs. placebo night) up to one month apart.
  Percent time asleep spent below an arterial oxygen saturation of 90% measured via pulse oximetry during overnight in-laboratory polysomnography.
Change in sleep efficiency (eszopiclone and lemborexant night vs. placebo night) | Two non-consecutive single night sleep studies (eszopiclone and lemborexant night vs. placebo night) up to one month apart.
  Percent time spent asleep divided by the recording time from lights out to lights on during overnight in-laboratory polysomnography
Change in arousal index (eszopiclone and lemborexant night vs. placebo night) | Two non-consecutive single night sleep studies (eszopiclone and lemborexant night vs. placebo night) up to one month apart.
  Number of cortical arousals per hour of sleep during overnight in-laboratory polysomnography.
Change in respiratory control (eszopiclone and lemborexant night vs. placebo night) | Two non-consecutive single night sleep studies (eszopiclone and lemborexant night vs. placebo night) up to one month apart.
  Loop gain and the ventilatory response to arousal (units: % eupnea) during overnight in-laboratory polysomnography.
Change in the respiratory arousal threshold (eszopiclone and lemborexant night vs. placebo night) | Two non-consecutive single night sleep studies (eszopiclone and lemborexant night vs. placebo night) up to one month apart.
  Threshold to arousal (units: % eupnea) during overnight in-laboratory polysomnography.
Change in airway collapsibility (eszopiclone and lemborexant night vs. placebo night) | Two non-consecutive single night sleep studies (eszopiclone and lemborexant night vs. placebo night) up to one month apart.
  Vpassive (units: % eupnea) during overnight in-laboratory polysomnography.
Change in pharyngeal muscle response (eszopiclone and lemborexant night vs. placebo night) | Two non-consecutive single night sleep studies (eszopiclone and lemborexant night vs. placebo night) up to one month apart.
  Vcompensation (units: % eupnea) during overnight in-laboratory polysomnography.
Baseline OSA endotype and whether they are associated with changes in OSA severity | Baseline sleep study
  Exploratory analysis to determine if baseline OSA endotypes as defined above (outcomes 7-10) are associated with changes in OSA severity as measured via the AHI- outcome 1 (eszopiclone and lemborexant night vs. placebo night)
Change in next morning balance (eszopiclone and lemborexant night vs. placebo night) | Next morning following two non-consecutive single night sleep studies (eszopiclone and lemborexant night vs. placebo night) up to one month apart.
  Stand on AMTI AccuSway Balance Board, eyes open and eyes closed 1 minute each. To evaluate balance in the next morning after eszopiclone and lemborexant night vs. placebo night (units: distance from center in cm)
Change in perceived sleepiness (eszopiclone and lemborexant night vs. placebo night) | Next morning following two non-consecutive single night sleep studies (eszopiclone and lemborexant night vs. placebo night) up to one month apart.
  Next day perceived sleepiness assessed via the Karolinska Sleepiness Scale (10 point scale where 1=extremely alert and 10=extremely sleepy)
Change in driving simulator performance (eszopiclone and lemborexant night vs. placebo night) | Next morning following two non-consecutive single night sleep studies (eszopiclone and lemborexant night vs. placebo night) up to one month apart.
  Next day alertness as measured via the Australian-developed (AusEd) driving simulator performance task (units: SD of steering deviation from median line).
Change in psycho-motor vigilance (eszopiclone and lemborexant night vs. placebo night) | Next morning following two non-consecutive single night sleep studies (eszopiclone and lemborexant night vs. placebo night) up to one month apart.
  Next day alertness as measured via the psychomotor vigilance test (PVT) (units m/s) higher values indicate worse performance.

CONTACTS AND LOCATIONS:
Overall Officials: Danny J Eckert, PhD, Principal Investigator — Flinders University
Locations (1):
- Flinders University, Adelaide Institute for Sleep Health, Bedford Park, South Australia, Australia

IPD SHARING:
Plan to Share IPD: Undecided
Our Participant Information Consent Form (PICF) asks if the participant is happy for their information to be shared with other researchers if it is deidentified. Deidentified individual participant data (IPD) might be made available to other researchers upon reasonable request and subject to ethical approval. Requests must include a methodologically sound proposal and will be reviewed by the Principal Investigator.

REFERENCES:
- [Background] Murphy P, Moline M, Mayleben D, Rosenberg R, Zammit G, Pinner K, Dhadda S, Hong Q, Giorgi L, Satlin A. Lemborexant, A Dual Orexin Receptor Antagonist (DORA) for the Treatment of Insomnia Disorder: Results From a Bayesian, Adaptive, Randomized, Double-Blind, Placebo-Controlled Study. J Clin Sleep Med. 2017 Nov 15;13(11):1289-1299. doi: 10.5664/jcsm.6800. PMID 29065953
- [Background] Terauchi M, Cheng JY, Yardley J, Pinner K, Moline M, Malhotra M, Inabe K, Nishida M, Pappadopulos E. Efficacy and safety of lemborexant in midlife women with insomnia disorder. Menopause. 2023 Aug 1;30(8):839-848. doi: 10.1097/GME.0000000000002209. Epub 2023 Jun 20. PMID 37339396
- [Background] Xue T, Wu X, Li J, Chen S, Wang Z, Tan X, Wang Z, Zhang J. Different doses of dual orexin receptor antagonists in primary insomnia: a Bayesian network analysis. Front Pharmacol. 2023 May 16;14:1175372. doi: 10.3389/fphar.2023.1175372. eCollection 2023. PMID 37261282
- [Background] Habiba U, Waseem R, Shaikh TG, Waseem S, Ahmed SH, Asghar MS. Correction to: Comparative efficacy and safety of lemborexant 5 mg versus 10 mg for the treatment of insomnia: a systematic review. Neurol Sci. 2023 May;44(5):1833. doi: 10.1007/s10072-023-06626-x. No abstract available. PMID 36650297
- [Background] Habiba U, Waseem R, Shaikh TG, Waseem S, Ahmed SH, Asghar MS. Comparative efficacy and safety of lemborexant 5 mg versus 10 mg for the treatment of insomnia: a systematic review. Neurol Sci. 2023 May;44(5):1533-1541. doi: 10.1007/s10072-023-06601-6. Epub 2023 Jan 12. PMID 36633778
- [Background] Cheng JY, Lorch D, Lowe AD, Uchimura N, Hall N, Shah D, Moline M. A randomized, double-blind, placebo-controlled, crossover study of respiratory safety of lemborexant in moderate to severe obstructive sleep apnea. J Clin Sleep Med. 2024 Jan 1;20(1):57-65. doi: 10.5664/jcsm.10788. PMID 37677076
- [Background] Cheng JY, Filippov G, Moline M, Zammit GK, Bsharat M, Hall N. Respiratory safety of lemborexant in healthy adult and elderly subjects with mild obstructive sleep apnea: A randomized, double-blind, placebo-controlled, crossover study. J Sleep Res. 2020 Aug;29(4):e13021. doi: 10.1111/jsr.13021. Epub 2020 Mar 18. PMID 32187781
- [Background] Eckert DJ, Malhotra A, Wellman A, White DP. Trazodone increases the respiratory arousal threshold in patients with obstructive sleep apnea and a low arousal threshold. Sleep. 2014 Apr 1;37(4):811-9. doi: 10.5665/sleep.3596. PMID 24899767
- [Background] Eckert DJ, Owens RL, Kehlmann GB, Wellman A, Rahangdale S, Yim-Yeh S, White DP, Malhotra A. Eszopiclone increases the respiratory arousal threshold and lowers the apnoea/hypopnoea index in obstructive sleep apnoea patients with a low arousal threshold. Clin Sci (Lond). 2011 Jun;120(12):505-14. doi: 10.1042/CS20100588. PMID 21269278
- [Background] Messineo L, Eckert DJ, Lim R, Chiang A, Azarbarzin A, Carter SG, Carberry JC. Zolpidem increases sleep efficiency and the respiratory arousal threshold without changing sleep apnoea severity and pharyngeal muscle activity. J Physiol. 2020 Oct;598(20):4681-4692. doi: 10.1113/JP280173. Epub 2020 Aug 30. PMID 32864734
- [Background] Messineo L, Carter SG, Taranto-Montemurro L, Chiang A, Vakulin A, Adams RJ, Carberry JC, Eckert DJ. Addition of zolpidem to combination therapy with atomoxetine-oxybutynin increases sleep efficiency and the respiratory arousal threshold in obstructive sleep apnoea: A randomized trial. Respirology. 2021 Sep;26(9):878-886. doi: 10.1111/resp.14110. Epub 2021 Jun 23. PMID 34164887
- [Background] Carter SG, Eckert DJ. Effects of hypnotics on obstructive sleep apnea endotypes and severity: Novel insights into pathophysiology and treatment. Sleep Med Rev. 2021 Aug;58:101492. doi: 10.1016/j.smrv.2021.101492. Epub 2021 Apr 22. PMID 33965721
- [Background] Carter SG, Carberry JC, Grunstein RR, Eckert DJ. Randomized Trial on the Effects of High-Dose Zopiclone on OSA Severity, Upper Airway Physiology, and Alertness. Chest. 2020 Jul;158(1):374-385. doi: 10.1016/j.chest.2020.02.057. Epub 2020 Mar 18. PMID 32197956
- [Background] Carter SG, Carberry JC, Cho G, Fisher LP, Rollo CM, Stevens DJ, D'Rozario AL, McKenzie DK, Grunstein RR, Eckert DJ. Effect of 1 month of zopiclone on obstructive sleep apnoea severity and symptoms: a randomised controlled trial. Eur Respir J. 2018 Jul 19;52(1):1800149. doi: 10.1183/13993003.00149-2018. Print 2018 Jul. PMID 29976648
- [Background] Carter SG, Berger MS, Carberry JC, Bilston LE, Butler JE, Tong BK, Martins RT, Fisher LP, McKenzie DK, Grunstein RR, Eckert DJ. Zopiclone Increases the Arousal Threshold without Impairing Genioglossus Activity in Obstructive Sleep Apnea. Sleep. 2016 Apr 1;39(4):757-66. doi: 10.5665/sleep.5622. PMID 26715227
- [Background] Edwards BA, Eckert DJ, McSharry DG, Sands SA, Desai A, Kehlmann G, Bakker JP, Genta PR, Owens RL, White DP, Wellman A, Malhotra A. Clinical predictors of the respiratory arousal threshold in patients with obstructive sleep apnea. Am J Respir Crit Care Med. 2014 Dec 1;190(11):1293-300. doi: 10.1164/rccm.201404-0718OC. PMID 25321848
- [Background] Eckert DJ. Phenotypic approaches to obstructive sleep apnoea - New pathways for targeted therapy. Sleep Med Rev. 2018 Feb;37:45-59. doi: 10.1016/j.smrv.2016.12.003. Epub 2016 Dec 18. PMID 28110857
- [Background] Gray EL, McKenzie DK, Eckert DJ. Obstructive Sleep Apnea without Obesity Is Common and Difficult to Treat: Evidence for a Distinct Pathophysiological Phenotype. J Clin Sleep Med. 2017 Jan 15;13(1):81-88. doi: 10.5664/jcsm.6394. PMID 27655455
- [Background] Zinchuk A, Edwards BA, Jeon S, Koo BB, Concato J, Sands S, Wellman A, Yaggi HK. Prevalence, Associated Clinical Features, and Impact on Continuous Positive Airway Pressure Use of a Low Respiratory Arousal Threshold Among Male United States Veterans With Obstructive Sleep Apnea. J Clin Sleep Med. 2018 May 15;14(5):809-817. doi: 10.5664/jcsm.7112. PMID 29734986
- [Background] Ghadiri M, Grunstein RR. Clinical side effects of continuous positive airway pressure in patients with obstructive sleep apnoea. Respirology. 2020 Jun;25(6):593-602. doi: 10.1111/resp.13808. Epub 2020 Mar 24. PMID 32212210
- [Background] Patil SP, Ayappa IA, Caples SM, Kimoff RJ, Patel SR, Harrod CG. Treatment of Adult Obstructive Sleep Apnea With Positive Airway Pressure: An American Academy of Sleep Medicine Systematic Review, Meta-Analysis, and GRADE Assessment. J Clin Sleep Med. 2019 Feb 15;15(2):301-334. doi: 10.5664/jcsm.7638. PMID 30736888
- [Background] Rotenberg BW, Murariu D, Pang KP. Trends in CPAP adherence over twenty years of data collection: a flattened curve. J Otolaryngol Head Neck Surg. 2016 Aug 19;45(1):43. doi: 10.1186/s40463-016-0156-0. PMID 27542595
- [Background] Baillieul S, Tamisier R, Eckert DJ, Pepin JL. Current Knowledge and Perspectives for Pharmacological Treatment in OSA. Arch Bronconeumol. 2022 Oct;58(10):681-684. doi: 10.1016/j.arbres.2021.12.013. Epub 2022 Jan 6. No abstract available. English, Spanish. PMID 35312500
- [Background] Eckert DJ, White DP, Jordan AS, Malhotra A, Wellman A. Defining phenotypic causes of obstructive sleep apnea. Identification of novel therapeutic targets. Am J Respir Crit Care Med. 2013 Oct 15;188(8):996-1004. doi: 10.1164/rccm.201303-0448OC. PMID 23721582
- [Background] Thomas E, Micic G, Adams R, Eckert DJ. Pharmacological management of co-morbid obstructive sleep apnoea and insomnia. Expert Opin Pharmacother. 2023 Sep-Dec;24(18):1963-1973. doi: 10.1080/14656566.2023.2292186. Epub 2024 Jan 5. PMID 38099435
- [Background] Sweetman A, Lack L, McEvoy RD, Antic NA, Smith S, Chai-Coetzer CL, Douglas J, O'Grady A, Dunn N, Robinson J, Paul D, Eckert D, Catcheside PG. Cognitive behavioural therapy for insomnia reduces sleep apnoea severity: a randomised controlled trial. ERJ Open Res. 2020 May 17;6(2):00161-2020. doi: 10.1183/23120541.00161-2020. eCollection 2020 Apr. PMID 32440518
- [Background] Benjafield AV, Ayas NT, Eastwood PR, Heinzer R, Ip MSM, Morrell MJ, Nunez CM, Patel SR, Penzel T, Pepin JL, Peppard PE, Sinha S, Tufik S, Valentine K, Malhotra A. Estimation of the global prevalence and burden of obstructive sleep apnoea: a literature-based analysis. Lancet Respir Med. 2019 Aug;7(8):687-698. doi: 10.1016/S2213-2600(19)30198-5. Epub 2019 Jul 9. PMID 31300334
- [Background] Sweetman A, Lack L, McEvoy RD, Smith S, Eckert DJ, Osman A, Carberry JC, Wallace D, Nguyen PD, Catcheside P. Bi-directional relationships between co-morbid insomnia and sleep apnea (COMISA). Sleep Med Rev. 2021 Dec;60:101519. doi: 10.1016/j.smrv.2021.101519. Epub 2021 Jun 23. PMID 34229295
- [Background] Meira E Cruz M, Kryger MH, Morin CM, Palombini L, Salles C, Gozal D. Comorbid Insomnia and Sleep Apnea: mechanisms and implications of an underrecognized and misinterpreted sleep disorder. Sleep Med. 2021 Aug;84:283-288. doi: 10.1016/j.sleep.2021.05.043. Epub 2021 Jun 8. PMID 34214960